CLINICAL TRIAL: NCT04064502
Title: Chronıc Ankle Instabılıty And Assocıated Factors
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Collaborators: Yeditepe University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YeditepeYUPTR
Record Dates: First submitted 2019-07-24; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-07

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic Ankle Instability; Cumberland Ankle Instability Tool; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- volunteers: 273 adult volunteers ranging from 18-78 years old
  Interventions: Diagnostic Test: CHRONIC ANKLE INSTABILITY AND ASSOCIATED FACTORS:

INTERVENTIONS:
Diagnostic Test: CHRONIC ANKLE INSTABILITY AND ASSOCIATED FACTORS: — Questionnaire including sociodemographic information, general medical condition, history of orthopedic surgery, pain intensity, and the number of painful areas of the foot.

SUMMARY:
The purpose of this study was to evaluate the prevalence of chronic ankle instability using the Cumberland Ankle Instability Tool (CAIT) and investigate the independent associated factors. The data was collected from adult volunteers by questionnaire including sociodemographic information, general medical condition, history of orthopedic surgery, pain intensity, and the number of painful areas of the foot.

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is a common condition encountered with persistent symptoms of giving way, pain, and weakness and recurrent risk, which may lead to functional insufficiency. The purpose of this study was to evaluate the prevalence of chronic ankle instability using the Cumberland Ankle Instability Tool (CAIT) and investigate the independent associated factors.

The data was collected from adult volunteers by questionnaire including sociodemographic information, general medical condition, history of orthopedic surgery, pain intensity, and the number of painful areas of the foot. 273 adult volunteers participated in the study, through face to face or online. Subjects are classified as having CAI with a CAIT score ≤27.

ELIGIBILITY:
Inclusion Criteria:

* being volunteer
* volunteers above 18 years old

Exclusion Criteria:

* history of acute ankle sprain
* acute ankle fracture
* receiving/having received physiotherapy and rehabilitation programs for foot and ankle problems
* within the last 6 months,history of foot, ankle, and/or knee surgery
* neuromuscular disorders
* disorders affecting balance
* diabetes mellitus complications

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The cross-sectional study group consisted of 273 adult volunteers, ranging from 18-78 years old, who were recruited via social media to maximize outreach and insure a diverse target group.
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
chronic ankle instability | 6 months
  Cumberland Ankle Instability Tool
  (CAIT) is a 9-item questionnaire generating a score from 0 to 30 for each ankle, in which 0 is the worst possible score, meaning severe instability, and 30 is the best possible score, meaning stability. The CAIT is considered a reliable instrument to distinguish between stable and unstable ankles, meanwhile, measuring the severity of functional ankle instability.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Şaylı, MD, Prof., Study Chair — Yeditepe University Hospital; Şule Demirbaş, Asst.Prof., Study Chair — editepe University, Faculty of Health Sciences, Deparment of Physiotherapy and Rehabilitation; Feryal Subaşı, PT, Prof., Study Chair — Yeditepe University, Faculty of Health Sciences, Deparment of Physiotherapy and Rehabilitation; Ebru Akbuğa, MSc, PT, Principal Investigator — Yeditepe University, Faculty of Health Sciences, Deparment of Physiotherapy and Rehabilitation; Elif Tuğçe Çil, MSc, PT, Principal Investigator — Yeditepe University, Faculty of Health Sciences, Deparment of Physiotherapy and Rehabilitation
Locations (1):
- Uğur Şaylı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes